CLINICAL TRIAL: NCT01082679
Title: Treatment for Opioid Dependent Offenders
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: University of Wisconsin, Milwaukee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2008-0242
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2019-05

CONDITIONS: Opioid Dependence
Keywords: opioid dependent; methadone; Suboxone; buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Methadone; Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- methadone via specialty care (Other)
  Interventions: Drug: Methadone
- Suboxone via specialty care (Other)
  Interventions: Drug: buprenorphine (Suboxone)
- Suboxone via primary care (Other)
  Interventions: Drug: buprenorphine (Suboxone)

INTERVENTIONS:
Drug: Methadone — daily for 12 months
  Arms: methadone via specialty care
Drug: buprenorphine (Suboxone) — daily for 12 months
  Arms: Suboxone via primary care; Suboxone via specialty care

SUMMARY:
This pilot study is examining the feasibility of a primary care and a specialist treatment (methadone clinic) model of treatment for 15 offenders who are part of two community supervision programs: Drug Court and the Treatment Alternative Program (TAP) in Dane County. The questions addressed by future larger studies based upon the current pilot-feasibility study will center around whether access to primary health care as opposed to more traditional methadone treatment services will improve the health and criminal justice outcomes for participants.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of opioid dependence
* opioid positive urine drug screen
* participation in local Drug Treatment Court or Treatment Alternative Program
* women of childbearing potential who have a negative screening urine pregnancy test and are willing to use appropriate birth control methods during the duration of the study

Exclusion Criteria:

* current alcohol or sedative dependence
* pregnancy
* women who are currently breast-feeding
* complex psychiatric co-morbidity (e.g. suicidality, psychosis)
* complex medical co-morbidity (e.g. major cardiovascular, renal, or gastrointestinal/hepatic disease)
* current pharmacotherapy with an agent which is contraindicated in combination with Suboxone or methadone according to drug labeling
* paralytic ileus, coronary artery disease or heart arrhythmia, recent head injury, obstructive sleep apnea, severe asthma or COPD, end-stage renal disease, or severe morbid obesity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Retention rate of participants in the study | 12 months
  This study is focused on Dane County Drug Treatment Court and Treatment Alternative Program participants.
  The study will determine feasibility of monitoring participants in primary care as opposed to the usual standard of specialty care.
  Feasibility of monitoring participants will be studied in terms of retention rate of participants in the study

CONTACTS AND LOCATIONS:
Overall Officials: Randy Brown, MD, PhD, Principal Investigator — University of Wisconsin - Madison, Department of Family Medicine
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

REFERENCES:
- [Result] Brown R, Gassman M, Hetzel S, Berger L. Community-based treatment for opioid dependent offenders: a pilot study. Am J Addict. 2013 Sep-Oct;22(5):500-2. doi: 10.1111/j.1521-0391.2013.12049.x. Epub 2013 Apr 3. PMID 23952897